CLINICAL TRIAL: NCT04040985
Title: A Prospective, Multi-Center, Non-Randomized, Safety and Efficacy Clinical Study of the LEGION™ Primary Knee System for Primary Total Knee Replacement in Subject With Degenerative Knee Disease
Brief Title: LEGION™ Primary Safety and Efficacy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: There is no regulatory or otherwise commitment to continue to follow up to the 10-year time point. The study data had met the primary objectives. After a business review, Smith+Nephew had decided to terminate the study prematurely.
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 10-K300-95301
Record Dates: First submitted 2019-07-18; First posted 2019-08-01 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-01

CONDITIONS: Osteo Arthritis Knee; Total Knee Replacement
Keywords: LEGION™ Primary; TKA; Osteoarthritis of Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LEGION™ Primary (Other): LEGION™ Primary Total Knee Arthroplasty (TKA)
  Interventions: Procedure: Total Knee Arthroplasty using LEGION™ Total Knee System

INTERVENTIONS:
Procedure: Total Knee Arthroplasty using LEGION™ Total Knee System — Primary Total Knee Arthroscopy using LEGION™ Total Knee System

SUMMARY:
This study will look at the health results of using the LEGION™ Primary Knee System over a period of ten (10) years. This type of surgery uses an artificial knee made of plastic and metal. This study will enter subjects who suffer from a variety of conditions that have caused at least one of their knees to become nonfunctional. You are being asked to participate in the study because you have significant problems with your knee(s) and your study surgeon has determined that your knee(s) must be surgically replaced to improve your condition. If you decided to participate in this study, you will be one of approximately one hundred thirty-eight (138) subjects in the study.

DETAILED DESCRIPTION:
This is a prospective, consecutive series, multi-center clinical study of the LEGION™ Total Knee System. The study design was selected to assess the safety and effectiveness profile of the LEGION™ Total Knee System in subjects with degenerative knee disease requiring primary total knee replacement.

Subjects meeting the entrance criteria specified in this protocol will be approached to participate in the study and enrolled sequentially. Any consenting subjects meeting the inclusion criteria are not to be excluded unless they do not consent to participate. A nonrandomized, consecutive series of up to 138 subjects will be enrolled at a maximum of 8 research sites, with an expectation of 18 subjects (up to a maximum of 28 subjects) to be enrolled at each site. When 138 subjects are enrolled from all sites, enrollment will be stopped, regardless of the number contributed from each site. Sites will be selected for participation in the study at the discretion of Smith & Nephew.

Follow-up clinical assessments will be at Operative/Discharge, 3 months, 1 year, 2 years, 3 years, 5 years, 7 years and 10 years. Each subject will receive a standard radiographic evaluation at discharge that will be used for baseline analysis. Additional radiographic analysis will be performed at Operative/Discharge, 3 months, 1 year, 2 years, 3 years, 5 years, 7 years and 10 years.

ELIGIBILITY:
Inclusion Criteria: Subjects must meet all of the inclusion criteria:

* Subject is a candidate for the LEGION™ Primary Knee System according to the instructions for use
* Subject is of legal age and skeletally mature
* Subject is willing to sign and date an ethics-approved consent form and participate in the study
* Subject is willing to be available for ten-year follow-up postoperatively.

Exclusion Criteria: Subjects must not meet any of the exclusion criteria:

* Subject with immunosuppressive disorders
* Subject has grossly insufficient femoral or tibial bone stock
* Subject has an active localized or systemic infection
* Subject is pregnant
* Subject psychological or neurological conditions that would impair the subject's ability or willingness to restrict activities or follow medical advice during the course of this study
* Subject is a prisoner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2009-09-09 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2020-12-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Orthopaedic Associates of Vero Beach, Vero Beach, Florida
  - Iowa Orthopaedic Center, Des Moines, Iowa
  - Louisville Bone & Joint Specialist, PSC, Louisville, Kentucky
  - University Hip and Knee Specialists, Monroe, New Jersey
  - University Orthopaedic Associates, LLC, Somerset, New Jersey

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: knees
Period: Overall Study
Arm/Group | LEGION™ Primary
Started | 128; 138 knees
Completed (At the time this study was terminated early by the Sponsor, there were 17 participants enrolled that did not completed their final study visit. These participants were not considered to have withdrawn or discontinued from the study.) | 69; 77 knees
Not Completed | 59; 61 knees

BASELINE CHARACTERISTICS:
Population: The Safety Population (SAF) used as the analysis population. The SAF was defined as all knees (or participants) enrolled into the study that were implanted with the study device. There were 10 participants with bilaterally enrolled knees.
Units Other Than Participants: knees
Arm/Group | LEGION™ Primary
Number analyzed (Participants) | 128
Number analyzed (knees) | 138
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (8.45)
Age, Customized [Count of Units; unit: knees] — Measurement evaluated by unit (knees)
  knees
    Age Group: ≤ 60 years | 34
    Age Group: > 60 years | 104
Sex: Female, Male [Count of Units; unit: knees] — Measurement evaluated by unit (knees)
  knees
    Female | 89
    Male | 49
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 128
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.1 (6.06)
Knee side implanted with device [Count of Units; unit: knees]
  Left | 69
  Right | 69

OUTCOME MEASURES:

1. Primary Outcome: Implant Survivorship Percentage
Description: Kaplan-Meier (KM) implant survivorship where survivorship defined as percentage of knees where no revision was required for any reason through 120 months
Time Frame: Postoperatively through 120 months
Population: The Safety Population (SAF) used as the analysis population. All knees (or participants) enrolled into the study that were implanted with the study device with available data at the time frame indicated.
Measure: Number (95% Confidence Interval); unit: percentage of knees
Units Other Than Participants: knees
Arm/Group | LEGION™ Primary
Number analyzed (Participants) | 69
Number analyzed (knees) | 77
percentage of knees | 96.9 [93.4 to 100.0]

2. Secondary Outcome: Knee Society Score (KSS) - Performance
Description: The Knee Society Score (KSS) performance outcome comprised information on objective knee indicators related to everyday activities. The Performance Score ranged from 0 to 100 with a higher score indicating a better outcome.
Time Frame: Preoperative, 3 months, 12 months, 24 months, 36 months, 60 months, 84 months, 120 months
Population: The Safety Population (SAF) used as the analysis population. All knees (or participants) enrolled into the study that were implanted with the study device with available data at the time frame indicated. Data for 11 knees at the preoperative time frame were not included because the data was collected prior to signing consent.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: knees
Arm/Group | LEGION™ Primary
Number analyzed (Participants) | 125
Number analyzed (knees) | 135
score on a scale
  Preoperative: number analyzed (Participants) | 119
  Preoperative: number analyzed (knees) | 127
  Preoperative | 40.9 (15.5)
  3 months | 84.5 (15.8)
  12 months: number analyzed (Participants) | 121
  12 months: number analyzed (knees) | 131
  12 months | 94.2 (10.0)
  24 months: number analyzed (Participants) | 109
  24 months: number analyzed (knees) | 119
  24 months | 95.1 (9.0)
  36 months: number analyzed (Participants) | 100
  36 months: number analyzed (knees) | 110
  36 months | 96.5 (5.8)
  60 months: number analyzed (Participants) | 89
  60 months: number analyzed (knees) | 99
  60 months | 97.4 (5.6)
  84 months: number analyzed (Participants) | 72
  84 months: number analyzed (knees) | 80
  84 months | 94.4 (10.0)
  120 months: number analyzed (Participants) | 59
  120 months: number analyzed (knees) | 66
  120 months | 98.0 (5.3)

3. Secondary Outcome: Knee Society Score (KSS) - Function
Description: The Knee Society Score (KSS) function outcome comprised information on functional knee indicators related to walking & standing, standard activities, advanced activities, and discretionary activities. The Function Score ranged from 0 to 100 with a higher score indicating a better outcome.
Time Frame: Preoperative, 3 months, 12 months, 24 months, 36 months, 60 months, 84 months, 120 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: knees
Arm/Group | LEGION™ Primary
Number analyzed (Participants) | 126
Number analyzed (knees) | 136
score on a scale
  Preoperative: number analyzed (Participants) | 118
  Preoperative: number analyzed (knees) | 127
  Preoperative | 53.8 (15.8)
  3 months | 73.1 (18.2)
  12 months: number analyzed (Participants) | 121
  12 months: number analyzed (knees) | 131
  12 months | 88.1 (14.8)
  24 months: number analyzed (Participants) | 109
  24 months: number analyzed (knees) | 119
  24 months | 91.0 (14.5)
  36 months: number analyzed (Participants) | 99
  36 months: number analyzed (knees) | 110
  36 months | 90.4 (16.7)
  60 months: number analyzed (Participants) | 91
  60 months: number analyzed (knees) | 101
  60 months | 93.4 (12.6)
  84 months: number analyzed (Participants) | 74
  84 months: number analyzed (knees) | 83
  84 months | 87.9 (16.1)
  120 months: number analyzed (Participants) | 62
  120 months: number analyzed (knees) | 69
  120 months | 89.3 (13.8)

4. Secondary Outcome: Knee Osteoarthritis Outcome Score (KOOS) - Pain
Description: The Knee Osteoarthritis Outcome Score (KOOS) Pain subscale used a Likert scale from 0 (No Problems) to 4 (Extreme Problems). Scores are transformed to a 0-100 scale, with 0 indicated a worse outcome and 100 representing a better outcome.
Time Frame: Preoperative, 3 months, 12 months, 24 months, 36 months, 60 months, 84 months, 120 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: knees
Arm/Group | LEGION™ Primary
Number analyzed (Participants) | 126
Number analyzed (knees) | 136
score on a scale
  Preoperative: number analyzed (Participants) | 119
  Preoperative: number analyzed (knees) | 127
  Preoperative | 43.0 (17.0)
  3 months | 72.4 (16.7)
  12 months: number analyzed (Participants) | 120
  12 months: number analyzed (knees) | 130
  12 months | 88.6 (13.9)
  24 months: number analyzed (Participants) | 109
  24 months: number analyzed (knees) | 119
  24 months | 90.9 (13.1)
  36 months: number analyzed (Participants) | 99
  36 months: number analyzed (knees) | 109
  36 months | 92.5 (10.2)
  60 months: number analyzed (Participants) | 92
  60 months: number analyzed (knees) | 102
  60 months | 94.2 (8.4)
  84 months: number analyzed (Participants) | 74
  84 months: number analyzed (knees) | 83
  84 months | 93.1 (11.9)
  120 months: number analyzed (Participants) | 67
  120 months: number analyzed (knees) | 74
  120 months | 95.7 (7.8)

5. Secondary Outcome: Knee Osteoarthritis Outcome Score (KOOS) - Symptom
Description: The Knee Osteoarthritis Outcome Score (KOOS) Symptom subscale used a Likert scale from 0 (No Problems) to 4 (Extreme Problems). Scores are transformed to a 0-100 scale, with 0 indicated a worse outcome and 100 representing a better outcome.
Time Frame: Preoperative, 3 months, 12 months, 24 months, 36 months, 60 months, 84 months, 120 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: knees
Arm/Group | LEGION™ Primary
Number analyzed (Participants) | 126
Number analyzed (knees) | 136
score on a scale
  Preoperative: number analyzed (Participants) | 119
  Preoperative: number analyzed (knees) | 127
  Preoperative | 46.6 (20.2)
  3 months | 68.5 (15.5)
  12 months: number analyzed (Participants) | 121
  12 months: number analyzed (knees) | 131
  12 months | 83.3 (11.6)
  24 months: number analyzed (Participants) | 109
  24 months: number analyzed (knees) | 119
  24 months | 85.9 (13.1)
  36 months: number analyzed (Participants) | 99
  36 months: number analyzed (knees) | 109
  36 months | 88.4 (11.2)
  60 months: number analyzed (Participants) | 92
  60 months: number analyzed (knees) | 102
  60 months | 89.1 (9.7)
  84 months: number analyzed (Participants) | 74
  84 months: number analyzed (knees) | 83
  84 months | 90.9 (9.5)
  120 months: number analyzed (Participants) | 68
  120 months: number analyzed (knees) | 75
  120 months | 91.9 (10.0)

6. Secondary Outcome: Knee Osteoarthritis Outcome Score (KOOS) - Function in Daily Living (ADL)
Description: The Knee Osteoarthritis Outcome Score (KOOS) Function in Daily Living (ADL) subscale used a Likert scale from 0 (No Problems) to 4 (Extreme Problems). Scores are transformed to a 0-100 scale, with 0 indicated a worse outcome and 100 representing a better outcome.
Time Frame: Preoperative, 3 months, 12 months, 24 months, 36 months, 60 months, 84 months, 120 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: knees
Arm/Group | LEGION™ Primary
Number analyzed (Participants) | 126
Number analyzed (knees) | 136
score on a scale
  Preoperative: number analyzed (Participants) | 119
  Preoperative: number analyzed (knees) | 127
  Preoperative | 46.4 (18.1)
  3 months | 77.5 (15.2)
  12 months: number analyzed (Participants) | 121
  12 months: number analyzed (knees) | 131
  12 months | 88.3 (11.4)
  24 months: number analyzed (Participants) | 108
  24 months: number analyzed (knees) | 118
  24 months | 90.1 (12.5)
  36 months: number analyzed (Participants) | 99
  36 months: number analyzed (knees) | 109
  36 months | 93.0 (9.5)
  60 months: number analyzed (Participants) | 92
  60 months: number analyzed (knees) | 102
  60 months | 92.4 (9.6)
  84 months: number analyzed (Participants) | 73
  84 months: number analyzed (knees) | 82
  84 months | 91.8 (12.2)
  120 months: number analyzed (Participants) | 67
  120 months: number analyzed (knees) | 74
  120 months | 92.2 (12.5)

7. Secondary Outcome: Knee Osteoarthritis Outcome Score (KOOS) - Sports and Recreational Activities
Description: The Knee Osteoarthritis Outcome Score (KOOS) Sports and Recreational Activities subscale used a Likert scale from 0 (No Problems) to 4 (Extreme Problems). Scores are transformed to a 0-100 scale, with 0 indicated a worse outcome and 100 representing a better outcome.
Time Frame: Preoperative, 3 months, 12 months, 24 months, 36 months, 60 months, 84 months, 120 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: knees
Arm/Group | LEGION™ Primary
Number analyzed (Participants) | 117
Number analyzed (knees) | 125
score on a scale
  Preoperative | 17.0 (23.4)
  3 months: number analyzed (Participants) | 112
  3 months: number analyzed (knees) | 121
  3 months | 49.1 (32.9)
  12 months: number analyzed (Participants) | 103
  12 months: number analyzed (knees) | 110
  12 months | 66.7 (28.4)
  24 months: number analyzed (Participants) | 96
  24 months: number analyzed (knees) | 105
  24 months | 67.5 (28.7)
  36 months: number analyzed (Participants) | 85
  36 months: number analyzed (knees) | 92
  36 months | 76.1 (27.9)
  60 months: number analyzed (Participants) | 77
  60 months: number analyzed (knees) | 83
  60 months | 71.0 (30.5)
  84 months: number analyzed (Participants) | 66
  84 months: number analyzed (knees) | 75
  84 months | 69.5 (32.5)
  120 months: number analyzed (Participants) | 52
  120 months: number analyzed (knees) | 56
  120 months | 71.3 (33.5)

8. Secondary Outcome: Knee Osteoarthritis Outcome Score (KOOS) - Quality of Life (QoL)
Description: The Knee Osteoarthritis Outcome Score (KOOS) Quality of Life (QoL) subscale used a Likert scale from 0 (No Problems) to 4 (Extreme Problems). Scores are transformed to a 0-100 scale, with 0 indicated a worse outcome and 100 representing a better outcome.
Time Frame: Preoperative, 3 months, 12 months, 24 months, 36 months, 60 months, 84 months, 120 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: knees
Arm/Group | LEGION™ Primary
Number analyzed (Participants) | 126
Number analyzed (knees) | 136
score on a scale
  Preoperative: number analyzed (Participants) | 119
  Preoperative: number analyzed (knees) | 127
  Preoperative | 17.6 (15.7)
  3 months | 56.4 (21.9)
  12 months: number analyzed (Participants) | 121
  12 months: number analyzed (knees) | 131
  12 months | 76.5 (20.0)
  24 months: number analyzed (Participants) | 108
  24 months: number analyzed (knees) | 118
  24 months | 78.8 (20.3)
  36 months: number analyzed (Participants) | 99
  36 months: number analyzed (knees) | 109
  36 months | 82.8 (18.4)
  60 months: number analyzed (Participants) | 91
  60 months: number analyzed (knees) | 101
  60 months | 84.3 (18.7)
  84 months: number analyzed (Participants) | 74
  84 months: number analyzed (knees) | 83
  84 months | 82.5 (19.5)
  120 months: number analyzed (Participants) | 67
  120 months: number analyzed (knees) | 74
  120 months | 85.9 (18.7)

9. Secondary Outcome: Radiographic Evaluation - Radiolucent Lines
Description: Performed weight bearing AP and lateral standard x-rays to identify knees with presence or absence of radiolucent lines categorized as:
  * Findings in Femoral Zone
  * Findings in Tibial Mediolateral (ML) Zone
  * Findings in Tibial Anteroposterior (AP) Zone
  * Findings in Patella Zone
  * No Radiolucent Lines Found
Time Frame: Discharge, 3 months, 1 year, 2 years, 3 years, 5 years, 7 years, 10 years
Population: as for outcome 1
Measure: Count of Units; unit: knees
Units Other Than Participants: knees
Arm/Group | LEGION™ Primary
Number analyzed (Participants) | 128
Number analyzed (knees) | 138
knees
  Discharge: Findings in Femoral Zone | 0
  Discharge: Findings in Tibial ML Zone | 0
  Discharge: Findings in Tibial AP Zone | 0
  Discharge: Findings in Patella Zone | 0
  Discharge: No Radiolucent Lines Found | 138
  3 months: number analyzed (Participants) | 126
  3 months: number analyzed (knees) | 136
  3 months: Findings in Femoral Zone | 1
  3 months: Findings in Tibial ML Zone | 0
  3 months: Findings in Tibial AP Zone | 1
  3 months: Findings in Patella Zone | 0
  3 months: No Radiolucent Lines Found | 134
  1 year: number analyzed (Participants) | 122
  1 year: number analyzed (knees) | 132
  1 year: Findings in Femoral Zone | 0
  1 year: Findings in Tibial ML Zone | 0
  1 year: Findings in Tibial AP Zone | 4
  1 year: Findings in Patella Zone | 0
  1 year: No Radiolucent Lines Found | 128
  2 years: number analyzed (Participants) | 109
  2 years: number analyzed (knees) | 119
  2 years: Findings in Femoral Zone | 1
  2 years: Findings in Tibial ML Zone | 2
  2 years: Findings in Tibial AP Zone | 4
  2 years: Findings in Patella Zone | 1
  2 years: No Radiolucent Lines Found | 111
  3 years: number analyzed (Participants) | 102
  3 years: number analyzed (knees) | 112
  3 years: Findings in Femoral Zone | 2
  3 years: Findings in Tibial ML Zone | 3
  3 years: Findings in Tibial AP Zone | 2
  3 years: Findings in Patella Zone | 1
  3 years: No Radiolucent Lines Found | 104
  5 years: number analyzed (Participants) | 93
  5 years: number analyzed (knees) | 103
  5 years: Findings in Femoral Zone | 2
  5 years: Findings in Tibial ML Zone | 2
  5 years: Findings in Tibial AP Zone | 2
  5 years: Findings in Patella Zone | 3
  5 years: No Radiolucent Lines Found | 94
  7 years: number analyzed (Participants) | 75
  7 years: number analyzed (knees) | 84
  7 years: Findings in Femoral Zone | 2
  7 years: Findings in Tibial ML Zone | 3
  7 years: Findings in Tibial AP Zone | 2
  7 years: Findings in Patella Zone | 3
  7 years: No Radiolucent Lines Found | 74
  10 years: number analyzed (Participants) | 69
  10 years: number analyzed (knees) | 76
  10 years: Findings in Femoral Zone | 0
  10 years: Findings in Tibial ML Zone | 0
  10 years: Findings in Tibial AP Zone | 0
  10 years: Findings in Patella Zone | 2
  10 years: No Radiolucent Lines Found | 74

10. Secondary Outcome: Radiographic Evaluation - Observed Periosteal Hypertrophy, Implant Loosening, Osteolysis or Subsidence
Description: Performed weight bearing AP and lateral standard x-rays to identify knees that observed periosteal hypertrophy, implant loosening, osteolysis or subsidence (Yes/No).
Time Frame: Discharge, 3 months, 1 year, 2 years, 3 years, 5 years, 7 years, 10 years
Population: as for outcome 1
Measure: Count of Units; unit: knees
Units Other Than Participants: knees
Arm/Group | LEGION™ Primary
Number analyzed (Participants) | 128
Number analyzed (knees) | 138
knees
  Discharge: Yes | 0
  Discharge: No | 138
  3 months: number analyzed (Participants) | 126
  3 months: number analyzed (knees) | 136
  3 months: Yes | 1
  3 months: No | 135
  1 year: number analyzed (Participants) | 122
  1 year: number analyzed (knees) | 132
  1 year: Yes | 0
  1 year: No | 132
  2 years: number analyzed (Participants) | 109
  2 years: number analyzed (knees) | 119
  2 years: Yes | 0
  2 years: No | 119
  3 years: number analyzed (Participants) | 102
  3 years: number analyzed (knees) | 112
  3 years: Yes | 0
  3 years: No | 112
  5 years: number analyzed (Participants) | 93
  5 years: number analyzed (knees) | 103
  5 years: Yes | 2
  5 years: No | 101
  7 years: number analyzed (Participants) | 75
  7 years: number analyzed (knees) | 84
  7 years: Yes | 2
  7 years: No | 82
  10 years: number analyzed (Participants) | 69
  10 years: number analyzed (knees) | 76
  10 years: Yes | 2
  10 years: No | 74

11. Secondary Outcome: Radiographic Evaluation - Observed Patellar Problem
Description: Performed weight bearing AP and lateral standard x-rays to identify knees that observed patellar problems (Yes/No).
Time Frame: Discharge, 3 months, 1 year, 2 years, 3 years, 5 years, 7 years, 10 years
Population: as for outcome 1
Measure: Count of Units; unit: knees
Units Other Than Participants: knees
Arm/Group | LEGION™ Primary
Number analyzed (Participants) | 128
Number analyzed (knees) | 138
knees
  Discharge: Yes | 0
  Discharge: No | 138
  3 months: number analyzed (Participants) | 126
  3 months: number analyzed (knees) | 136
  3 months: Yes | 0
  3 months: No | 136
  1 year: number analyzed (Participants) | 122
  1 year: number analyzed (knees) | 132
  1 year: Yes | 0
  1 year: No | 132
  2 years: number analyzed (Participants) | 109
  2 years: number analyzed (knees) | 119
  2 years: Yes | 1
  2 years: No | 118
  3 years: number analyzed (Participants) | 102
  3 years: number analyzed (knees) | 112
  3 years: Yes | 3
  3 years: No | 109
  5 years: number analyzed (Participants) | 93
  5 years: number analyzed (knees) | 103
  5 years: Yes | 0
  5 years: No | 103
  7 years: number analyzed (Participants) | 75
  7 years: number analyzed (knees) | 84
  7 years: Yes | 1
  7 years: No | 83
  10 years: number analyzed (Participants) | 69
  10 years: number analyzed (knees) | 76
  10 years: Yes | 0
  10 years: No | 76

ADVERSE EVENTS:
Time Frame: Adverse events were collected from surgery up to 10 years.
Description: Device-related Adverse Event (AE) were any related to device use (e.g., component breakage). All postoperative device & surgery related AEs were reported. Specifically, all component removals (and/or revisions) whether device-related or not were recorded. Other AEs were classified as device-related/non device-related based on their frequency, medical significance, & circumstance. Thus, Investigators reported AE relatedness for device & procedure in the same Case Report Form (CRF) question.
Arm/Group | LEGION™ Primary
All-Cause Mortality (participants affected / at risk) | 4/128
Serious Adverse Events (participants affected / at risk) | 75/128
Other Adverse Events (participants affected / at risk) | 116/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEGION™ Primary (N=128)
Anemic (Metabolism and nutrition disorders) | 1 (1) — Unrelated
Ankle fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Back surgery, due to lumbar spondylosis (Musculoskeletal and connective tissue disorders) | 3 (3) — Unrelated
Buttock abcess (Infections and infestations) | 1 (1) — Unrelated
Cardiac stent for heart disease, bigemy (Cardiac disorders) | 1 (1) — Unrelated
Chronic rotator cuff tear (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Compression fracture, lower back, due to degeneration lumbar disc (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Compression fracture, lower back (Musculoskeletal and connective tissue disorders) | 2 (2) — Unrelated
Compression fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Death - cardiac event (Cardiac disorders) | 1 (1) — Unrelated
Death - Parkinson's Disease (Nervous system disorders) | 1 (1) — Unrelated
Death - Unknown cause (General disorders) | 2 (2) — Unrelated
Deep vein thrombosis, calf (Vascular disorders) | 1 (1) — Procedure Related
Deep vein thrombosis, lower extremity (Vascular disorders) | 1 (1) — Procedure Related
Deep vein thrombosis, popliteal vein (Vascular disorders) | 1 (1) — Procedure Related
Deep vein thrombosis (Vascular disorders) | 1 (2) — Procedure Related
Deep vein thrombosis (Vascular disorders) | 1 (1) — Unrelated
Diabetes Mellitus (Metabolism and nutrition disorders) | 2 (2) — Unrelated
Erosive esophagitis (Gastrointestinal disorders) | 1 (1) — Unrelated
Foot navicular stress fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Fracture after component insertion and cementing (Injury, poisoning and procedural complications) | 1 (1) — Device Related
Hip fracture with bipolar hemiarthroplasty and knee contusion (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Hip osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4) — Unrelated
Hip pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Hyperparathyroidism (Endocrine disorders) | 1 (1) — Unrelated
Hypertension (Cardiac disorders) | 1 (1) — Unrelated
Hypotension (Cardiac disorders) | 1 (1) — Procedure Related
Hypotension (Cardiac disorders) | 1 (1) — Unrelated
Infected total knee (Injury, poisoning and procedural complications) | 2 (2) — Device Related
Infection (Infections and infestations) | 1 (1) — Procedure Related
Knee arthrofibrosis (Musculoskeletal and connective tissue disorders) | 2 (2) — Procedure Related
Knee effusion (Musculoskeletal and connective tissue disorders) | 1 (1) — Device Related
Knee lateral retinacular release (Surgical and medical procedures) | 1 (1) — Device + Procedure Related
Knee manipulation under anesthesia, due to arthrofibrosis (Musculoskeletal and connective tissue disorders) | 1 (1) — Device + Procedure Related
Knee manipulation under anesthesia, due to stiffness (Musculoskeletal and connective tissue disorders) | 3 (3) — Procedure Related
Knee manipulation under anesthesia (Surgical and medical procedures) | 1 (1) — Device Related
Knee manipulation under anesthesia (Surgical and medical procedures) | 2 (2) — Procedure Related
Knee osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) — Unrelated
Knee patellar tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) — Procedure Related
Knee stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) — Procedure Related
Lap band procedure (Surgical and medical procedures) | 1 (1) — Unrelated
Leg swelling (General disorders) | 1 (1) — Procedure Related
Lung cancer, stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Unrelated
Mechanical loosening of internal knee patella button (Product Issues) | 1 (1) — Device Related
Myocardial infarction (Cardiac disorders) | 1 (1) — Procedure Related
Olecranon and distal radius fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Patellar clunking (Product Issues) | 1 (1) — Device Related
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Unrelated
Radial head fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Respiratory failure, altered mental status and atelactasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Procedure Related
Shoulder arthoscopy, due to torn rotator cuff (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Spine and ribs fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Splenic artery aneurism embolisation (Vascular disorders) | 1 (1) — Unrelated
Superficial wound debricence, post-op (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated
Total hip arthroplasty, due to hip pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Total hip arthroplasty, due to osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) — Unrelated
Total hip arthroplasty (Surgical and medical procedures) | 1 (1) — Unrelated
Total knee arthroplasty, due to knee pain secondary to degenerative joint disease (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Total knee arthroplasty, due to knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Total knee arthroplasty, due to osteoarthritis (Musculoskeletal and connective tissue disorders) | 8 (8) — Unrelated
Total knee arthroplasty (Surgical and medical procedures) | 11 (11) — Unrelated
Urinary retention (Renal and urinary disorders) | 1 (1) — Unrelated
Vertebral compression fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Wrist fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEGION™ Primary (N=128)
Achilles tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Anemia (Metabolism and nutrition disorders) | 2 (2) — Unrelated
Ankle sprain (Musculoskeletal and connective tissue disorders) | 2 (2) — Unrelated
Ankle swelling (Musculoskeletal and connective tissue disorders) | 1 (1) — Device + Procedure Related
Back and hip pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Back pain and SI joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) — Unrelated
Bakers cyst (Musculoskeletal and connective tissue disorders) | 1 (1) — Procedure Related
Bladder control loss and pain (Renal and urinary disorders) | 1 (1) — Unrelated
Blisters near incision (Skin and subcutaneous tissue disorders) | 1 (1) — Procedure Related
Carpal tunnel, bilateral (Nervous system disorders) | 1 (1) — Unrelated
Chronic venous insufficiency lower extremities, bilateral (Vascular disorders) | 1 (1) — Unrelated
Clicking knee (Musculoskeletal and connective tissue disorders) | 2 (2) — Device + Procedure Related
Clicking knee (Musculoskeletal and connective tissue disorders) | 1 (1) — Device Related
Constipation (Gastrointestinal disorders) | 2 (2) — Unrelated
Contusion, due to fall (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated
Cyst anterior knee (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Unrelated
Degeneration of lumbar intervertebral disc and spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (2) — Unrelated
Diarrhea (Gastrointestinal disorders) | 1 (1) — Unrelated
Distal fibular avulsion and left wrist injury, due to fall (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Dizziness (General disorders) | 1 (1) — Unrelated
Dupuytren's middle finger (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Erythema of incision (Skin and subcutaneous tissue disorders) | 1 (1) — Procedure Related
Exostosis lateral femoral condyle knee (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Fall (General disorders) | 3 (3) — Unrelated
Fever (General disorders) | 3 (4) — Unrelated
Finger contusions (Skin and subcutaneous tissue disorders) | 1 (2) — Unrelated
Foot and ankle pain (Musculoskeletal and connective tissue disorders) | 2 (2) — Unrelated
Foot and ankle partial tear (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Foot neuropathy (Nervous system disorders) | 1 (1) — Unrelated
Foot pain, bilateral (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Foot pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Hand pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Headache (General disorders) | 1 (2) — Unrelated
Heretopic ossification (Musculoskeletal and connective tissue disorders) | 1 (1) — Device Related
Herniated disc (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Heterotopic ossification infra patella (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Heterotopic ossification of femoral component (Musculoskeletal and connective tissue disorders) | 1 (1) — Device + Procedure Related
Heterotopic ossification (Musculoskeletal and connective tissue disorders) | 1 (1) — Device Related
Hip and knee pain, due to IT band friction syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Hip pain and sciatica (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Hip pain, bilateral (Musculoskeletal and connective tissue disorders) | 2 (2) — Unrelated
Hip pain, due to osteoarthritis and trochanteric bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Hip pain, due to osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Hip pain, lateral (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Hip pain (Musculoskeletal and connective tissue disorders) | 3 (5) — Unrelated
Hypertrophic scar formation (Skin and subcutaneous tissue disorders) | 1 (1) — Procedure Related
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) — Unrelated
Index finder (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Index finger (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
IT band irritation (Musculoskeletal and connective tissue disorders) | 1 (1) — Procedure Related
Knee arthrofibrosis (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Knee bakers cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Procedure Related
Knee buckling (Musculoskeletal and connective tissue disorders) | 2 (2) — Unrelated
Knee clicking and grinding (Musculoskeletal and connective tissue disorders) | 1 (1) — Device + Procedure Related
Knee clicking (Musculoskeletal and connective tissue disorders) | 3 (3) — Device + Procedure Related
Knee clicking (Musculoskeletal and connective tissue disorders) | 5 (6) — Device Related
Knee contusion, bilateral (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated
Knee contusion, due to fall (Skin and subcutaneous tissue disorders) | 4 (4) — Unrelated
Knee contusion (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated
Knee crackling when standing (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Knee hematoma and contusion, due to fall (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated
Knee hematoma (Skin and subcutaneous tissue disorders) | 1 (1) — Procedure Related
Knee hyperextension (Musculoskeletal and connective tissue disorders) | 1 (1) — Device + Procedure Related
Knee instability (Musculoskeletal and connective tissue disorders) | 1 (1) — Procedure Related
Knee instability (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Knee lateral swelling (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Knee lump and pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Knee osteoarthritis with crepitus (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Knee osteoarthritis (Musculoskeletal and connective tissue disorders) | 8 (8) — Unrelated
Knee pain and bruising, due to fall (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated
Knee pain with swelling and redness around patella (Skin and subcutaneous tissue disorders) | 1 (1) — Procedure Related
Knee pain, bilateral (Musculoskeletal and connective tissue disorders) | 1 (2) — Unrelated
Knee pain, due to contusion (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated
Knee pain, due to fall (Musculoskeletal and connective tissue disorders) | 1 (1) — Device + Procedure Related
Knee pain, due to fall (Musculoskeletal and connective tissue disorders) | 6 (6) — Unrelated
Knee pain, due to MVA (Musculoskeletal and connective tissue disorders) | 1 (1) — Device Related
Knee pain, due to osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (11) — Unrelated
Knee pain (Musculoskeletal and connective tissue disorders) | 4 (4) — Device + Procedure Related
Knee pain (Musculoskeletal and connective tissue disorders) | 2 (2) — Device Related
Knee pain (Musculoskeletal and connective tissue disorders) | 3 (3) — Procedure Related
Knee pain (Musculoskeletal and connective tissue disorders) | 13 (15) — Unrelated
Knee pes anserine bursitis (Musculoskeletal and connective tissue disorders) | 2 (2) — Unrelated
Knee popping (Musculoskeletal and connective tissue disorders) | 1 (1) — Device + Procedure Related
Knee popping (Musculoskeletal and connective tissue disorders) | 1 (1) — Procedure Related
Knee posteriolateral popping, occasional (Musculoskeletal and connective tissue disorders) | 1 (1) — Procedure Related
Knee soft tissue pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Knee stiffness post manipulation (Musculoskeletal and connective tissue disorders) | 1 (1) — Procedure Related
Knee stiffness, post op (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Knee stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Knee strain (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Knee swelling, due to infection (Infections and infestations) | 1 (1) — Procedure Related
Knee swelling, intermittent (Musculoskeletal and connective tissue disorders) | 1 (1) — Procedure Related
Knee swelling (Musculoskeletal and connective tissue disorders) | 1 (1) — Procedure Related
Knee swelling (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Knee tenderness along MCL (Musculoskeletal and connective tissue disorders) | 1 (1) — Procedure Related
Knee tenderness along MCL (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Knee tenderness and bruising, due to fall (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated
Knee tightness (Musculoskeletal and connective tissue disorders) | 1 (1) — Device + Procedure Related
Knee wound infection drainage (Infections and infestations) | 1 (1) — Procedure Related
Lateral knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Lateral patella tilt and impingment (Musculoskeletal and connective tissue disorders) | 1 (1) — Device Related
Lateral subluxation and patella tilt (Musculoskeletal and connective tissue disorders) | 1 (2) — Device Related
Leg pain, due to advanced arthritic changes of lumbar spine (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Leg swelling and ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) — Procedure Related
Lower back and groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Lower back and hip pain (Musculoskeletal and connective tissue disorders) | 2 (2) — Unrelated
Lower back pain and sciatica (Nervous system disorders) | 1 (1) — Unrelated
Lower back pain radiating to lower extremities (Nervous system disorders) | 1 (1) — Unrelated
Lower back pain with radiculopathy (Nervous system disorders) | 1 (1) — Unrelated
Lower back pain, due to degeneration of lumbar intervertebral disc, spondylosis (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Lower back pain (Musculoskeletal and connective tissue disorders) | 5 (5) — Unrelated
Lower calf clot (Vascular disorders) | 1 (1) — Unrelated
Lower extremity swelling (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated
Lumbar pain, due to sciatica-lumbar radiculopathy (Nervous system disorders) | 1 (1) — Unrelated
Lumbar radiculitis and spasm (Nervous system disorders) | 1 (1) — Unrelated
Lumbar radiculopathy and sciatica (Nervous system disorders) | 1 (1) — Unrelated
Lumbar spondylosis (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
MVA (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Patella heterotopic ossification (Musculoskeletal and connective tissue disorders) | 1 (1) — Device Related
Patella periosteal hypertrophy (Musculoskeletal and connective tissue disorders) | 1 (1) — Device Related
Patellar Subluxation (Musculoskeletal and connective tissue disorders) | 1 (1) — Device + Procedure Related
Peroneal nerve palsy (Nervous system disorders) | 1 (1) — Procedure Related
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Reabsorption on the medial tibial plateau (Musculoskeletal and connective tissue disorders) | 1 (1) — Device Related
Sacroilliac pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Sciatica and spasm (Nervous system disorders) | 1 (2) — Unrelated
Sciatica (Nervous system disorders) | 1 (1) — Unrelated
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unrelated
Shoulder bursitis and osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Shoulder fracture, due to fall (Musculoskeletal and connective tissue disorders) | 2 (2) — Unrelated
Shoulder pain, bilateral (Musculoskeletal and connective tissue disorders) | 2 (2) — Unrelated
Shoulder pain, due to impingement (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Shoulder pain, due to severe glenohumeral DJD (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Shoulder pain (Musculoskeletal and connective tissue disorders) | 5 (9) — Unrelated
Shoulder rotator cuff tear (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Shoulder stiffness, due to post op (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Shuffling gait (General disorders) | 1 (1) — Unrelated
Spinal stenosis and sciatica (General disorders) | 1 (1) — Unrelated
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 (6) — Unrelated
Spondylosis and allied disorder (Musculoskeletal and connective tissue disorders) | 1 (4) — Unrelated
Spondylosis and sacroilliac joint inflamed (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Stenosing tenosynovitis finger (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Thumb pain, due to arthritis (Musculoskeletal and connective tissue disorders) | 1 (2) — Unrelated
Tingling anterior thigh (Nervous system disorders) | 1 (1) — Unrelated
Total hip, post-op (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Total shoulder, pre op (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Trochanteric bursitis (Musculoskeletal and connective tissue disorders) | 2 (2) — Unrelated
Urinary tract infection (Renal and urinary disorders) | 3 (3) — Unrelated
Vertigo (Nervous system disorders) | 1 (1) — Unrelated
Weakness, due to low sodium (Metabolism and nutrition disorders) | 1 (1) — Unrelated
Weight gain (General disorders) | 1 (1) — Unrelated

LIMITATIONS AND CAVEATS:
Limitations of study included high drop-out rate, which was additionally influenced by impact COVID-19 had on subject retention & follow-up rate. Participants lost to follow-up based on presumed loss of power at the 7-year (62.7% follow-up rate) & 10-year (58.5%) time points led to early study termination by Sponsor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2011-02-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT04040985/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/85/NCT04040985/SAP_001.pdf